CLINICAL TRIAL: NCT05397327
Title: Virtual 3D Surgical Planning for Tibial Plateau Fractures: A Multicenter Prospective Randomized Controlled Trial
Brief Title: 3D Virtual Planning for Tibial Plateau Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other); Flinders Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NL2022-13629
Record Dates: First submitted 2022-05-10; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Tibial Plateau Fracture
MeSH Terms: conditions — Tibial Plateau Fractures

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional planning group (No Intervention): Conventional preoperative planning using x-rays and 2D and 3D CT scan
- 3D virtual planning group (Experimental): Preoperative planning using x-rays, 2D and 3D CT scans and 3D virtual planning software
  Interventions: Other: 3D virtual planning software

INTERVENTIONS:
Other: 3D virtual planning software — 3D virtual planning software developed by Sectra AB (Linköping, Sweden)
  Arms: 3D virtual planning group

SUMMARY:
Tibial plateau fractures are often complex fractures and need a good preoperative planning. The investigators think that a 3D virtual planning software will help the surgeons to get a better understanding of the fracture and therefore want to study the value of 3D virtual planning software in the preoperative planning of tibial plateau fractures. The investigators hypothesize that this software will shorten the duration of surgery, decrease the peroperative bloodloss and the number of complications.

Patients with tibial plateau fractures who need surgical treatment will be asked to participate in this study. After participants have given informed consent, they will be randomized between a 'traditional preoperative planning' and a '3D virtual preoperative planning' group. Surgeons will plan their surgery using traditional planning tools (X-rays and CT scan) or traditional planning tools ánd the 3D virtual planning software.

6 weeks, 3 months and 6 months after surgery, participants will be asked to fill in 2 questionnaires about knee pain and knee function. After surgery a CT scan or X-ray will be performed conform standard of care in the hospital.

DETAILED DESCRIPTION:
Patients with tibial plateau fractures are traditionally challenging to treat, especially the complex fracture patterns in which anatomic reconstruction of the articular surface can be very demanding. In a previous study, the researchteam showed that surgical decision-making should be guided by recognition of specific fracture characteristics, rather than the 'classic' classification of fractures by Schatzker. Recognition of these specific tibial plateau fracture patterns has been proven reliable and reproducible to guide surgeons plan their approach, reduction techniques and fixation.

Building on our improved understanding of (complex) tibial plateau fracture patterns, and how these specific fracture characteristics guide our surgical management, the next step includes meticulous pre-operative surgical planning to achieve the best functional results for our patients. A new state-of-the-art tool is currently available to aid surgeons in 3D virtual planning of approach, reduction strategy, and even application of hardware (i.e. size of plates and lengths of screws (https://sectra.com/medical/product/sectra-3d-trauma/).

Recent studies on virtual surgical planning for fracture care have shown variable results. One study concluded that there was a significant reduction in duration of surgery in about 75.0% of all cases. Another study showed improvement of the outcomes of acetabular fracture surgery by reduced duration of the surgery and improved quality of the reduction. However, a third study showed that 3D virtual reality is inferior compared to 3D printed models on acetabular fractures in terms of interobserver agreement. In conclusion, the added value of virtual preoperative planning has yet to be determined.

If virtual surgical planning is as promising as some of the previous results show, it could also have a significant impact on the surgical reduction in the treatment of tibial plateau fractures. This might lead to a reduction of duration of surgery, less complications and better patient related outcomes, such as postoperative pain and knee function.

Therefore, the investigators would like to compare the conventional preoperative planning with the preoperative planning with use of the virtual planning software of Sectra AB for tibial plateau fractures in terms of duration of surgery, surgical complications and patient related outcomes.

To see if the virtual planning software is comparable with the postoperative situation, the investigators would like to compare the preoperative virtual plan with the postoperative CT scan in terms of residual displacement and placement of the osteosynthesis material.

Primary Objective:

What is the added value of pre-operative virtual 3D surgical planning compared to traditional pre-surgical planning (i.e. surgeons' interpretation and written planning of standard 2D- and 3D CT-imaging) in patients with tibial plateau fractures in terms of duration of surgery?

Secondary Objective(s):

What is the added value of pre-operative virtual 3D surgical planning compared to traditional pre-surgical planning (i.e. surgeons' interpretation and written planning of standard 2D- and 3D CT-imaging) in patients with tibial plateau fractures in terms of

* postoperative complications?
* peroperative deviations of surgical planning?
* quality of post-operative reduction (i.e. reduction of step-off)?
* patient related outcomes (i.e. postoperative pain and knee function)?

For this study, the investigators have chosen to perform a randomized controlled trial to reduce the risk of selection bias. Participants will be divided in two groups, where in the conventional group trauma surgeons will plan their surgery using X-rays, 2D and 3D CT scans. In the virtual group, surgeons will plan their surgery using the virtual 3D planning software of Sectra AB and X-rays, 2D and 3D CT scans.

In both groups, surgery will be performed conform standard of care. This means that the preoperative planning is used as a guideline for the surgery and there will be deviated from the planning if deemed necessary for the surgery.

Postoperative, surgeons will be asked to fill in questionnaires to determine deviations of the preoperative plan, time spent planning and satisfaction. Patients will be asked to fill in questionnaires to determine functional outcome and health related quality of life, a postoperative CT scan will be performed after surgery to determine quality of postoperative reduction, according to our standard-of-care.

Quality of reduction on a CT or X-ray does not always match with patient experienced outcomes. Therefore, the investigators have chosen to not only measure quality of reduction, but also patient related outcomes, such as postoperative knee function and health related quality of life. Because of this possible mismatch, the investigators have chosen for reduction of operation time as our primary outcome. A longer operation time is associated with more postoperative surgical complications and blood loss. Furthermore, operation time is valuable and therefore expensive. A reduction in operation time would therefore not only have an effect on patient related outcomes, but also have effect on healthcare costs.

This study will take place at the following three level I trauma centers:

* Flinders University Medical Center, Adelaide, Australia
* Radboud University Medical Center, Nijmegen, the Netherlands
* Massachusetts General Hospital, Boston, United States of America

The investigators will ask patients who present themselves at the emergency department with a tibial plateau fracture that needs surgical treatment within 14 days of the injury to participate in this study. If they are willing to participate, an informed consent will be signed and furthermore, they will receive an information folder with specified information about this research study.

Surgical residents and surgeons will be informed about this study through an e-mail with a short outline of the research. They will be asked to inform the researcher when there is a patient with a tibial plateau fracture who needs surgical treatment. The researcher will visit the emergency department or ward to inform the patient and sign the informed consent. A patient can give informed consent until two days before the planned surgery to ensure the trauma surgeon has enough time to plan the surgery thoroughly.

When included, patients will randomly be divided into two groups through sealed opaque envelopes:

* Group 1: preoperative planning using the 3D virtual planning software of SECTRA
* Group 2: traditional preoperative planning (i.e. surgeons' interpretation and written planning of standard 2D- and 3D CT-imaging).

Concealed randomization will be obtained with the randomizer.org software and stratified by centers.

Per trauma center, the investigators will train three experienced trauma surgeons in using the SECTRA 3D virtual planning software. These surgeons perform the majority (i.e. 95%) of all patients admitted with tibial plateau fractures. The investigators will ask the surgeons from both the traditional and virtual planning groups to keep track of time they spent planning the surgery. After planning the surgery, the surgeons will fill in a questionnaire where they indicate their surgical plan (i.e. which screws and plates they are planning to use and which surgical approach they attend to perform) and time spent planning.

After the surgery, the surgeons will fill in a questionnaire where they will indicate if they deviated from the pre-operative plan and if they are satisfied with the postoperative result. Using the operative notes, the investigators will determine the used screws, plates and surgical approach and the total duration of surgery.

Postoperative patients will get a CT-scan to determine the quality of the postoperative reduction. After 6 weeks, 12 weeks and 6 months the investigators will determine functional outcome and health related quality of life using the 'Knee injury and Osteoarthritis Score' (KOOS) questionnaire, and the Short Form - 36 (SF-36) questionnaire.

The investigators will use CastorEDC for creating the patient and surgeon questionnaires and for storing patient information at the secured digital research environment of Radboud University Medical Center. All patient and surgeon information will be pseudonymized by the department of Radiology and Nuclear Medicine of the participating hospital, therefore subjects privacy is protected. This key will be deleted after data collection is finished. For analysis, these questionnaires will be exported to SPSS. The data of the statistical analysis and the results will also be stored at the secured digital research environment. The data will be kept for 15 years. Only researchers involved in the study have access to the data.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients of 18 years or older with a tibial plateau fracture who will receive surgical treatment for this fracture

Exclusion Criteria:

* patients with (general) bone diseases or osseous malformation syndromes,
* ipsilateral limb fractures,
* complicated tibial plateau fractures that need an external fixator,
* previous tibial plateau fractures
* previous surgical treatment of the tibial plateau

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Duration of surgery | Intraoperative
  Time in minutes from start of surgery till end of surgery

SECONDARY OUTCOMES:
Blood loss | Intraoperative
  Amount of blood loss in milliliters during surgery
Surgical complications | up to 30 days postoperative
  Number of complications related to performed surgery or to condition
Perioperative deviations | Immediately after x-ray or CT scan is performed
  Number of perioperative deviations of the perioperative plan
Quality of reduction | Immediately after x-ray or CT scan is performed
  Postoperative step off in millimeters as measured on postoperative CT scan or X-ray
Quality of reduction | Immediately after x-ray or CT scan is performed
  Postoperative gap in millimeters as measured on postoperative CT scan or X-ray
Postoperative knee function | Measured at 6 weeks, 3 months and 6 months postoperative
  Participant indicated postoperative knee function as measured with the KOOS questionnaire (score between 0 and 100, with 100 being no pain/restrictions in knee function) and SF-36 questionnaire (score between 0 and 100, with 100 being no limitations in social functioning)
Postoperative knee pain | Measured at 6 weeks, 3 months and 6 months postoperative
  Participant indicated postoperative knee function as measured with the KOOS questionnaire (score between 0 and 100, with 100 being no pain/restrictions in knee function) and SF-36 questionnaire (score between 0 and 100, with 100 being no limitations in social functioning)

CONTACTS AND LOCATIONS:
Overall Officials: Job Doornberg, Professor, Principal Investigator — University Medical Center Groningen
Locations (3):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Flinders Medical Center, Adelaide, South Australia, Australia
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will use the digital research environment (DRE), developed by a collaboration of hospitals in the Netherlands, to share anonymized individual participant data between the three participating centers.
  Participant data that will be shared is:
  * 3D Virtual planning software
  * Time spent planning
  * Fracture Characteristics
  * Surgeon satisfaction
  * Patient Demographics
    * Age
    * Sex
    * Mechanism of injury
    * Comorbidities
    * BMI
    * Duration of surgery
    * Number of complications
    * Perioperative deviations
    * Quality of reduction
    * Knee pain and function
  * Surgeon characteristics
    * Area of practice
    * Sex
    * Specialization
    * Years in practice
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after inclusion of the first patient. The data will be vailable until 6 months after inclusion of the last patient
Access Criteria: Only the research team will have access to the data
URL: https://mydre.org/